CLINICAL TRIAL: NCT02634515
Title: A Randomized, Single-center, Double-blind, 2-period Crossover, Euglycemic Glucose Clamp Study in Healthy Subjects to Demonstrate PK and PD Equivalence of Julphar Insulin R and Huminsulin® Normal
Brief Title: Pharmacokinetic (PK) Bioequivalence and Pharmacodynamics of Julphar Insulin R and Huminsulin® Normal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Julphar Gulf Pharmaceutical Industries (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry); Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: INSULCT001
Record Dates: First submitted 2015-12-11; First posted 2015-12-18 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes Mellitus
Keywords: soluble human insulin, biosimilar
MeSH Terms: conditions — Diabetes Mellitus | interventions — Biosimilar Pharmaceuticals

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Julphar Insulin R (Experimental): Julphar Insulin R, soluble human insulin, biosimilar, 100 IU/mL, single subcutaneous injection of 0.3 IU/kg body weight
  Interventions: Drug: Julphar Insulin R (soluble human insulin, biosimilar)
- Huminsulin® Normal (Active Comparator): Huminsulin® Normal, soluble human insulin, reference, 100 IU/mL, single subcutaneous injection of 0.3 IU/kg body weight
  Interventions: Drug: Huminsulin® Normal (soluble human insulin, reference)

INTERVENTIONS:
Drug: Julphar Insulin R (soluble human insulin, biosimilar) — investigational insulin, Julphar Insulin R (soluble human insulin)
  Other Names: Julphar Insulin R
  Arms: Julphar Insulin R
Drug: Huminsulin® Normal (soluble human insulin, reference) — marketed product, Huminsulin® Normal (soluble human insulin
  Other Names: Huminsulin® Normal
  Arms: Huminsulin® Normal

SUMMARY:
This study in healthy volunteers aimed to demonstrate similar PK and PD properties of the new short-acting human soluble insulin, Julphar Insulin R, and the already approved reference insulin, Huminsulin® Normal. The trial participants received both study treatments on two separate dosing days.

DETAILED DESCRIPTION:
The daily injection of insulin is a necessity for many patients with diabetes mellitus in order to treat hyperglycemia. Julphar Insulin R and Huminsulin® Normal are both soluble insulins intended for subcutaneous administration and consist of a neutral solution containing recombinant human insulin as the active ingredient. The new insulin, Julphar Insulin R is biosimilar to Huminsulin® Normal. Demonstration of bioequivalence from a PK and PD perspective of the two insulins are necessary to achieve market approval for Julphar Insulin R.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject).
* Healthy male or female subjects.
* Age between 18 and 55 years, both inclusive.
* Body Mass Index (BMI) between 18.5 and 28.0 kg/m^2, both inclusive.
* Fasting plasma glucose (FPG) ≤5.6 mmol/L (100 mg/dL).

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products.
* Receipt of any IMP within 3 months prior to screening.
* Any history or presence of a life threatening disease (i.e., cancer except basal cell skin cancer or squamous cell skin cancer), or of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, haematological, neurological, musculoskeletal, articular, psychiatric, systemic, ocular, gynaecologic (females), or infectious disease, or signs of acute illness as judged by the Investigator.
* Surgery within 12 weeks before the start of the study or blood donation of more than 500 mL (or considerable blood loss) or plasma donation within the last 3 months.
* Increased risk of thrombosis, e.g., subjects with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator.
* Haemoglobin < 8.0 mmol/L (male) or < 6.4 mmol/L (female), total leukocyte count < 3.0 x 10^9/L, thrombocytes < 100 x 10^9/L, serum creatinine levels ≥ 126 µmol/L (male) or ≥ 111 µmol/L (female), alanine aminotransferase (ALT) > 2 x the upper limit of normal (ULN), bilirubin > 3 x ULN, alkaline phosphatase > 2 x ULN.
* Supine blood pressure (BP) at screening (after resting for 5 minutes in a supine position) outside the range of 90 to 140 mmHg for systolic BP or 50 to 90 mmHg for diastolic BP (excluding white-coat hypertension; therefore, if a repeated measurement shows values within the range, the subject can be included in the trial) and/or resting supine pulse < 50 beats per minute.
* Clinically significant abnormal standard 12-lead ECG after 5 minutes resting in a supine position at screening, as judged by the Investigator.
* Any disease or condition that, in the opinion of the Investigator, would represent an unacceptable risk for the subject's safety.
* Subject known to be positive for Hepatitis Bs antigen (HBsAg) or Hepatitis C antibodies (or diagnosed with active hepatitis according to local practice) or test positive at screening for human immunodeficiency virus Type 1 (HIV-1) antibodies, HIV Type 2 (HIV 2) antibodies, or HIV-1 antigen according to locally used diagnostic testing.
* History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol.
* Any medication (prescription and non-prescription drugs) within 14 days before first trial drug administration, with the exception of stable treatment with thyroid hormones, paracetamol for occasional use to treat pain, and if female, with the exception of hormonal contraception or menopausal hormone replacement therapy.
* Significant history of alcoholism or drug/chemical abuse as per Investigator's judgement or a positive result in the urine drug/alcohol screen at the screening visit or consuming more than 21 units of alcohol per week (1 unit of alcohol equals approximately 330 mL of beer, 1 glass of wine (120 mL), or 40 mL spirits).
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day) who is not able or willing to refrain from smoking and use of nicotine substitute products 1 day before and during the inpatient period/trial.
* Subject with mental incapacity or language barriers precluding adequate understanding or cooperation or who, in the opinion of the Investigator or their general practitioner, should not participate in the trial.
* Potentially noncompliant or uncooperative during the trial, as judged by the Investigator.
* Female who is pregnant, breast feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods (adequate contraceptive measures are defined as surgical sterilisation, implants, injectables, combined oral contraceptives, hormonal intrauterine device, sexual abstinence, or vasectomised partner).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
PK: AUCins.0-12h, area under the serum insulin concentration time curve from 0 to 12 hours | 12 hours
  primary endpoint according EMA guideline
PK: Cins.max, maximum serum insulin concentration | 12 hours
  primary endpoint according EMA guideline
PD: AUCGIR.0-last, area under the glucose infusion rate curve from 0 hours until the end of the glucose clamp | 12 hours
  primary endpoint according EMA guideline
PD: GIRmax, maximum glucose infusion rate | 12 hours
  primary endpoint according EMA guideline

SECONDARY OUTCOMES:
PK: AUCins.0-4h,area under the serum insulin concentration time curve from 0 to 4 hours | 4 hours
PK: AUCins.0-6h,area under the serum insulin concentration time curve from 0 to 6 hours | 6 hours
PK: AUCins.6-12h, area under the serum insulin concentration time curve from 6 to 12 hours | 12 hours
PK: AUCins.0-infinity, area under the serum insulin concentration time curve from 0 (dosing) to infinity | 12 hours
PK: tmax, time to maximum serum insulin concentration | 12 hours
PK: t50%-early, time to serum insulin increased to 50%, respectively of maximum serum insulin concentration | 12 hours
PK: t50%-late, time to serum insulin decreased to 50%, respectively of maximum serum insulin concentration | 12 hours
PK: t½, terminal serum elimination half-life calculated as t½=ln2/λz | 12 hours
PK: λz, terminal elimination rate constant of insulin | 12 hours
PK: MRT, mean residence time | 12 hours
PK: CL/F, total body clearance | 12 hours
PK: V/F, volume of distribution | 12 hours
PD: AUCGIR0-4h, AUCGIR0-6h, AUCGIR6-last, areas under the glucose infusion rate curve in the indicated time-intervals | 12 hours
PD: tGIRmax, time to maximum glucose infusion rate curve | 12 hours
PD: tGIR50%-early, time to GIR increased to 50%, respectively of maximum GIR value | 12 hours
PD: tGIR50%-late, time to GIR decreased to 50%, respectively of maximum GIR value | 12 hours
PD: onset of action - time from trial product administration until blood glucose concentration has decreased at least 0.3 mmol/L (5 mg/dL) from baseline | 12 hours
  baseline is defined as the mean of blood glucose levels measured with Super GL analyser at -6, -4,and -2 minutes before trial product administration
Adverse events | from first trial drug administration until final examination (up to 30 days for each patient)
Hypoglycaemic events | from first trial drug administration until the final examination (up to 30 days for each patient)
Physical examination findings | from screening until the final examination (up to 58 days for each patient)
Vital signs recordings | from screening until the final examination (up to 58 days for each patient)
Electrocardiograms | from screening until the final examination(up to 58 days for each patient)
Laboratory safety variables (haematology, biochemistry, and urinalysis) | from screening until the final examination (up to 58 days for each patient)
Assessment of local tolerability at the injection site | from first trial drug administration until the final examination (up to 58 days for each patient)
  The local tolerability at the injection site will be evaluated by means of the following assessments:
  * Spontaneous pain
  * Pain on palpation
  * Itching
  * Erythema
  * Oedema
  * Induration Each of these assessments will be reported on a scale of 0 (none), 1 (mild), 2 (moderate), and 3 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Hövelmann, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany